CLINICAL TRIAL: NCT06532071
Title: Advanced Imaging for Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Caravan (Other)
Responsible Party: Sponsor-Investigator, Peter Caravan, Professor of Radiology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P001746
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Pulmonary Fibrosis (Experimental): Participants with non-idiopathic pulmonary fibrosis interstitial lung disease (non-IPF ILD) will receive [68Ga]CBP8 and undergo PET combined with dynamic contrast-enhanced MRI
  Interventions: Drug: [68Ga]CBP8; Drug: Gadoterate Meglumine

INTERVENTIONS:
Drug: [68Ga]CBP8 — Participants will receive a single intravenous injection of up to 350 MBq of [68Ga]CBP8
Drug: Gadoterate Meglumine — Participants will receive a single intravenous injection of 0.05 mmol/kg gadoterate meglumine during DCE-MRI
  Other Names: Dotarem

SUMMARY:
The purpose of this study is to determine if measurements of active collagen deposition using [68Ga]CBP8 positron emission tomography (PET) and tissue injury using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) can predict an individual patient's pace of disease progression in non-idiopathic pulmonary fibrosis interstitial lung disease (non-IPF ILD) and identify which individuals will develop progressive pulmonary fibrosis.

DETAILED DESCRIPTION:
60 participants with non-idiopathic pulmonary fibrosis interstitial lung disease (non-IPF ILD) on stable dose immunosuppression treatment will be enrolled. Participants will undergo combined [68Ga]CBP8 positron emission tomography (PET) and dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) at baseline. The investigators will compare the ability of PET and MRI measurements performed over the whole lung and within regions of interest to identify participants who subsequently develop progressive pulmonary fibrosis as determined by changes in pulmonary function testing, quantitative fibrosis on high-resolution computed tomography, and respiratory symptoms over 24 months. The investigators will also test whether combining the PET and MRI measurements results in more accurate prediction of progression than either modality alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 with a diagnosis of chronic hypersensitivity pneumonitis, connective tissue-associated ILD (due to rheumatoid arthritis, systemic sclerosis, mixed connective tissue disease), or undifferentiated ILD.
2. On stable dose immunosuppression treatment (with prednisone, mycophenolate mofetil, and/or rituximab) for at least 3 months.
3. Pulmonary fibrosis, defined as honeycombing, traction bronchiectasis, or reticular opacities on HRCT performed within 1 year to or at Visit 1.
4. FVC of >/= 45% and DLCO >/= 25% predicted on PFTs performed at Visit 1.

Exclusion Criteria:

1. Current or prior exposure to FDA approved anti-fibrotic therapy.
2. Extent of emphysema greater than extent of fibrosis.
3. Pregnancy or plans to become pregnant at baseline or during follow-up.
4. Contraindications to MRI.
5. Contraindications to receiving gadolinium-based contrast agents.
6. Research-related radiation exposure exceeds 50 mSv in the prior year.
7. Estimated glomerular filtration rate (eGFR) < 30 mL/min (only for individuals with a history of chronic kidney disease).
8. Clinically significant PH defined by use of pulmonary vasodilatory therapy.
9. Respiratory infection within the prior 6 weeks.
10. Smoking of any kind within the prior 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of progressive pulmonary fibrosis | Up to 24 months
  Defined by the 2022 ATS guideline definition of progressive pulmonary fibrosis (PPF) which defines PPF as satisfying 2 of 3 criteria within 12 months: worsening symptoms, physiologic progression (absolute decline in FVC ≥ 5% or absolute decline in DLCO ≥ 10%), or radiologic evidence of disease progression.

SECONDARY OUTCOMES:
Decline of forced vital capacity (FVC) ≥ 5% from baseline | Up to 24 months
  FVC will be measured at baseline, 6, 12, 18, and 24 months
Decline of forced vital capacity (FVC) ≥10% from baseline | Up to 24 months
  FVC will be measured at baseline, 6, 12, 18, and 24 months
Decline of diffusing capacity for carbon monoxide (DLCO) ≥15% from baseline | Up to 24 months
  DLCO will be measured at baseline, 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Montesi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Izquierdo-Garcia D, Desogere P, Fur ML, Shuvaev S, Zhou IY, Ramsay I, Lanuti M, Catalano OA, Catana C, Caravan P, Montesi SB. Biodistribution, Dosimetry, and Pharmacokinetics of 68Ga-CBP8: A Type I Collagen-Targeted PET Probe. J Nucl Med. 2023 May;64(5):775-781. doi: 10.2967/jnumed.122.264530. Epub 2022 Dec 8. PMID 37116909
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537